CLINICAL TRIAL: NCT02334891
Title: Kyoto Congestive Heart Failure Study
Acronym: KCHF
Status: Completed | Type: Observational
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University, Graduate School of Medicine
Other Study IDs: E2311
Record Dates: First submitted 2014-12-28; First posted 2015-01-08 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Congestive Heart Failure; Heart Failure, Diastolic; Heart Failure, Systolic; Elderly Frail; Guideline Adherence
Keywords: congestive heart failure; heart failure, diastolic; heart failure, systolic; elderly frail; guideline adherence
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Standard — Standard management

SUMMARY:
The purpose of this study is to investigate the patient characteristics, selection of treatment, and factors associated with clinical outcomes in Japanese patients with acutely decompensated congestive heart failure.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) has been markedly increasing in Japan due to the rapid aging of the society and the Westernization of lifestyle that facilitates the development of coronary artery disease. The prognosis of patients with CHF still remains poor, despite the recent advances in medical and surgical treatment. Elderly heart failure patients with preserved ejection and multiple comorbidity may account for significant portion among CHF patients in the real world clinical practice, however; most of previous prospective cohort studies excluded these patients. The KCHF registry, an all-comer, prospective, multicenter registry, was designed to investigate all patients who admitted to the hospital due to acutly decompensated CHF. The aim of this study was to clarify the patients characteristics , selection of treatment, and prognosis of patients with acutly decompensated CHF in the real-world clinical practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

* All patients who admitted to the participating centers due to acutly decompensated CHF defined by modified Framingham criteria
* Patients who underwent heart failure treatment including intravenus drug

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who admitted to the participating centers due to acutly decompensated CHF defined by modified Framingham criteria
Sampling Method: Non-Probability Sample
Enrollment: 4056 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
hospital mortality | 1-year

SECONDARY OUTCOMES:
functional level at discharge measured by NYHA classification | 1-year
improvement of dyspnea level at discharge measured by Likert scale | 1-year
walking ability at discharge categorized by ambulatory, wheelchair (outdoor only), wheelchair (outdoor and indoor), bedridden | 1-year
any severe ventricular arrhythmic event during hospitalization | 1-year
onset of atrial fibrillation events during hospitalization | 1-year
any bradyarrhythmic event during hospitalization | 1-year
any stroke during hospitalization | 1-year
any cardiac surgery during hospitalization | 1-year
any cateter intervention during hospitalization | 1-year
any device implantation during hospitalization | 1-year
bleeding events during hospitalization (GUSTO definition; moderate to severe) | 1-year
adverse drug events during hospitalization | 1-year
infectious diseases during hospitalization | 1-year
change of BNP at discharge (≧30% compared to BNP at admission ) | 1-year
worsening renal function at discharge (raise of Cr≧0.3mg/dl compared to Cr at admission ) | 1-year
usage of guideline recommended medicine during hospitalization | 1-year
usage of tolvaptan during hospitalization | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School and Faculty of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Kyoto University Hospital, Kyoto, Japan

REFERENCES:
- [Derived] Nishikawa R, Kato T, Morimoto T, Yaku H, Inuzuka Y, Tamaki Y, Yamamoto E, Ozasa N, Tada T, Sakamoto H, Seko Y, Shiba M, Yoshikawa Y, Yamashita Y, Kitai T, Taniguchi R, Iguchi M, Nagao K, Kawai T, Komasa A, Kawase Y, Morinaga T, Toyofuku M, Furukawa Y, Ando K, Kadota K, Sato Y, Kuwahara K, Kimura T; KCHF Study Investigators. The characteristics and outcomes in patients with acute heart failure who used tolvaptan: from KCHF registry. ESC Heart Fail. 2023 Oct;10(5):3141-3151. doi: 10.1002/ehf2.14494. Epub 2023 Aug 29. PMID 37644779
- [Derived] Aida K, Nagao K, Kato T, Yaku H, Morimoto T, Inuzuka Y, Tamaki Y, Yamamoto E, Yoshikawa Y, Kitai T, Taniguchi R, Iguchi M, Kato M, Takahashi M, Jinnai T, Kawai T, Komasa A, Nishikawa R, Kawase Y, Morinaga T, Su K, Kawato M, Seko Y, Inada T, Inoko M, Toyofuku M, Furukawa Y, Nakagawa Y, Ando K, Kadota K, Shizuta S, Ono K, Sato Y, Kuwahara K, Ozasa N, Kimura T. Prognostic Value of the Severity of Clinical Congestion in Patients Hospitalized for Decompensated Heart Failure: Findings From the Japanese KCHF Registry. J Card Fail. 2023 Aug;29(8):1150-1162. doi: 10.1016/j.cardfail.2023.01.003. Epub 2023 Jan 21. PMID 36690136
- [Derived] Nishimoto Y, Kato T, Morimoto T, Taniguchi R, Yaku H, Inuzuka Y, Tamaki Y, Yamamoto E, Yoshikawa Y, Kitai T, Iguchi M, Kato M, Takahashi M, Jinnai T, Ikeda T, Nagao K, Kawai T, Komasa A, Nishikawa R, Kawase Y, Morinaga T, Su K, Kawato M, Seko Y, Inoko M, Toyofuku M, Furukawa Y, Nakagawa Y, Ando K, Kadota K, Shizuta S, Ono K, Kuwahara K, Ozasa N, Sato Y, Kimura T. Public assistance in patients with acute heart failure: a report from the KCHF registry. ESC Heart Fail. 2022 Jun;9(3):1920-1930. doi: 10.1002/ehf2.13898. Epub 2022 Mar 15. PMID 35289117
- [Derived] Seko Y, Kato T, Morimoto T, Yaku H, Inuzuka Y, Tamaki Y, Ozasa N, Shiba M, Yamamoto E, Yoshikawa Y, Yamashita Y, Kitai T, Taniguchi R, Iguchi M, Nagao K, Jinnai T, Komasa A, Nishikawa R, Kawase Y, Morinaga T, Toyofuku M, Furukawa Y, Ando K, Kadota K, Sato Y, Kuwahara K, Kimura T; KCHF Study Investigators. Newly Diagnosed Infection After Admission for Acute Heart Failure: From the KCHF Registry. J Am Heart Assoc. 2021 Nov 16;10(22):e023256. doi: 10.1161/JAHA.121.023256. Epub 2021 Nov 3. PMID 34730004
- [Derived] Washida K, Kato T, Ozasa N, Morimoto T, Yaku H, Inuzuka Y, Tamaki Y, Seko Y, Yamamoto E, Yoshikawa Y, Kitai T, Yamashita Y, Iguchi M, Nagao K, Kawase Y, Morinaga T, Toyofuku M, Furukawa Y, Ando K, Kadota K, Sato Y, Kuwahara K, Kimura T. Risk Factors and Clinical Outcomes of Nonhome Discharge in Patients With Acute Decompensated Heart Failure: An Observational Study. J Am Heart Assoc. 2021 Aug 3;10(15):e020292. doi: 10.1161/JAHA.120.020292. Epub 2021 Jul 30. PMID 34325523
- [Derived] Nishimoto Y, Kato T, Morimoto T, Yaku H, Inuzuka Y, Tamaki Y, Yamamoto E, Yoshikawa Y, Kitai T, Taniguchi R, Iguchi M, Kato M, Takahashi M, Jinnai T, Ikeda T, Nagao K, Kawai T, Komasa A, Nishikawa R, Kawase Y, Morinaga T, Su K, Kawato M, Seko Y, Inoko M, Toyofuku M, Furukawa Y, Nakagawa Y, Ando K, Kadota K, Shizuta S, Ono K, Kuwahara K, Ozasa N, Sato Y, Kimura T. C-reactive protein at discharge and 1-year mortality in hospitalised patients with acute decompensated heart failure: an observational study. BMJ Open. 2020 Dec 29;10(12):e041068. doi: 10.1136/bmjopen-2020-041068. PMID 33376169
- [Derived] Yaku H, Kato T, Morimoto T, Inuzuka Y, Tamaki Y, Ozasa N, Yamamoto E, Yoshikawa Y, Kitai T, Kato M, Ikeda T, Furukawa Y, Nakagawa Y, Sato Y, Kuwahara K, Kimura T. Risk factors and clinical outcomes of functional decline during hospitalisation in very old patients with acute decompensated heart failure: an observational study. BMJ Open. 2020 Feb 16;10(2):e032674. doi: 10.1136/bmjopen-2019-032674. PMID 32066601